CLINICAL TRIAL: NCT04124341
Title: Prefrontal Cortical Stimulation (PCS) for Severe Treatment Resistant Depression
Brief Title: PCS in Severe Treatment Resistant Depression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PSYCH-2019-27331
Record Dates: First submitted 2019-10-10; First posted 2019-10-11 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Treatment Resistant Depression
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Prefrontal Cortical Stimulation (PCS) (Experimental): Stereotactically implanted bilateral PCS
  Interventions: Device: Prefrontal Cortical Stimulation (PCS)

INTERVENTIONS:
Device: Prefrontal Cortical Stimulation (PCS) — Prior to surgery, subjects will undergo a high resolution structural scan to identify anatomical landmarks for rostral anterior and lateral prefrontal cortex. Following identification of target areas, PCS quad leads will be projected over the anterior and lateral prefrontal cortex. Subjects will be kept in the hospital for a minimum of 72 hours for observation during which the investigators will obtain a high resolution spiral CT scan without contrast to confirm lead placements post-operatively and rule out any intra-cranial bleeds. Patients will receive analgesics which they may continue as an outpatient on as needed basis. During this 2-3 weeks recovery period, the attention to pain control and mood is critical. The research team will contact patients at least twice per week to check on their status.

SUMMARY:
This research study is designed to test if electrical stimulation of the surface of the brain in the frontal region will help treat depressive symptoms. Participants receive intermittent electrical stimulation to the brain, which involves surgically placing electric leads in between the tough fibrous membrane covering the surface of the brain and the surface of the brain itself. This type of stimulation is referred to as bilateral subdural prefrontal cortical stimulation (PCS) because it will specifically target the outer layer of the brain at the midline, right behind the forehead. It uses a pacemaker-like device, the Proclaim Elite SCS System (non-rechargeable) or the Eterna SCS System (rechargeable), both by Abbott Laboratories for stimulation.

Although the U.S. Food and Drug Administration (FDA) has approved the Proclaim Elite SCS system for brain stimulation for patients with chronic pain and muscular diseases, such as Parkinson's, its use is still investigational, and the surgery is still experimental for patients who have depression.

DETAILED DESCRIPTION:
This study has five distinct stages.

Stage 1: Baseline Assessments There is a 14-day baseline period to determine eligibility, including medical history, physical and neurological examinations, and medical test including EKG, blood work, pregnancy test, depression assessments and cognitive assessments. An MRI will also be done prior to implant in order to help the surgeon determine where best to place the leads.

Stage 2: Surgery If deemed to be medically eligible, participants will be hospitalized for a minimum of 3 days, during which they will undergo surgery to implant the device and leads. There will be testing of the leads to explore optimal testing parameters. According to the surgeon's judgment, participants may or may not receive stimulation for 3 weeks following surgery.

Stage 3: Acute phase (19 weeks) Following implantation, participants undergo a CT scan to ensure proper implantation. Later, participants complete 10 follow up visits where assessments of symptoms will be made. Additionally, the first visit will consist of the investigator programming the stimulator while participants watch various photographs with different emotional content and have their brain electrical activity recorded. This will help the investigator choose the best settings for treatment. Pregnancy tests will be done as appropriate.

Stage 4: Follow up (7 months) All participants who complete stage 3 will be offered continued treatment. Participants complete 7 monthly follow-up visits where assessments of symptoms are made. Pregnancy tests will be done as appropriate.

Stage 5: Long Term Follow up (4 years) All participants who complete stage 4 will be offered continued treatment. Participants complete follow up visits every three months, alternating between in person and over zoom. Assessments of symptoms are made. Pregnancy tests will be done as appropriate.

Objectives To demonstrate that PCS causes meaningful and sustained antidepressant response.

To demonstrate that precision functional mapping can identify individualized depression patterns which will lead to personalized maps for targeting the stimulation for an individual.

To establish safe parameters for PCS that do not generate after discharge seizures.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be able to provide written informed consent.
* Participant has a diagnosis of chronic (greater than or equal to 2 years) depressive episode as defined by DSM V criteria
* Participant has not had an adequate response to four or more adequate antidepressant treatments from at least two different antidepressant treatment categories in the current depressive episode according to the Antidepressant Treatment History Form (ATHF)
* Participant must have had ECT (Electroconvulsive Therapy) or refused to undergo ECT if clinically indicated to them
* Participant must have HRSD greater than or equal to 20 at study entry
* Participant must be able to complete the evaluations needed for this study including the functional imaging scans and the EEG Bayesian optimization sessions
* Participant must be under the care of a licensed psychiatrist, undergoing regular care evaluations, and inform study team of any change to care team during study participation
* Participant must agree to allow all forms of communication between investigators and study staff and any health care provider (current or having provided service within two years of enrollment)
* Participant must provide name and contact information for at least two people greater than or equal to 22 in age who reside within a 30 minute drive of the participant's residents and whom staff may contact as necessary during study participation
* Participant must be enrolled in a Medicare program

Exclusion Criteria:

* The PCS would (in the investigator's judgment) pose an unacceptable surgical or medical risk for the participant
* Participant is unable to undergo required full body magnetic resonance imaging (MRI) during the clinical study
* Participant is judged by the investigator to be acutely suicidal (e.g. within the 30 days prior to the PCS implant the participant has made a suicide attempt or gesture or has made specific plans or preparation to commit suicide or scores 21 or higher on the MSSI)
* In addition to the acute suicidal risks mentioned above, participant meets any of the following:

  1. Has made a suicide attempt within the previous 12 months that required medical treatment
  2. Has made greater than or equal to two suicide attempts in the past 12 months
  3. Has a clear-cut plan for suicide that states that she/he cannot guarantee that she/he will call her/his regular psychiatrist or the Investigator if the impulse to implement the plan becomes substantial during the study
  4. Is likely to attempt suicide within the next six months, in the Investigator's opinion
* Participant has a history of schizophrenia, schizoaffective disorder, or other psychotic disorder, or a current major depressive episode that includes psychotic features (commonly referred to as psychotic depression) according to the DSM V criteria
* Participant with a diagnosis of dementia with a Mini-Mental State Exam (MMSE) less than or equal to 23
* Participant with a positive urine pregnancy test
* Participant with a positive urine drug screen
* Participant with DBS (Deep Brain Stimulator)
* Participant with VNS (Vagus Nerve Stimulator) if the device was active in the last 6 months prior to study enrollment
* Participant with history of seizures
* Participant determined by surgical safety committee to have cerebral atrophy, neurodegenerative or neurovascular disease due to age or medical condition that would prohibit optimal surgical safety, per clinical MRI

Ages: 22 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2021-09-29 (Actual); Primary Completion 2031-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in HRSD Scores | 12 months
  Determine clinical change in depressive symptoms over first year of treatment

SECONDARY OUTCOMES:
Change in HRSD Scores | 60 months
  Determine whether clinical effects seen within the first year persist, improve, or worsen during an extended period of time

CONTACTS AND LOCATIONS:
Overall Officials: Ziad Nahas, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No